CLINICAL TRIAL: NCT03543098
Title: STaR (Surgical Timing and Rehabilitation) Trial for Multiple Ligament Knee Injuries
Brief Title: STaR Trial: Multiple Ligament Knee Injuries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Rhode Island Hospital (Other); Hospital for Special Surgery, New York (Other); Mayo Clinic (Other); New York University (Other); University of Cincinnati (Other); University of Kentucky (Other); University of Maryland (Other); University of Michigan (Other); University of Minnesota (Other); University of Missouri-Columbia (Other); University of New Mexico (Other); University of Washington (Other); Washington University School of Medicine (Other); San Antonio Military Medical Center (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); William Beaumont Army Medical Center (U.S. Federal Agency); TRIA Orthopaedic Center (Other); Wake Forest University (Other); Unity Health Toronto (Other); Western University, Canada (Other); Ochsner Health System (Other); Yale University (Other); OrthoCarolina Research Institute, Inc. (Other); Louisiana State University Health Sciences Center Shreveport (Other); Duke University (Other); University of Calgary (Other); Oregon Health and Science University (Other); Wake Forest University Health Sciences (Other); Orlando Health, Inc. (Other); Fraser Orthopaedic Institute (Unknown)
Responsible Party: Principal Investigator, James J. Irrgang, Professor and Chair, Department of Physical Therapy, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20110374; W81XWH-17-2-0073 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2018-05-08; First posted 2018-06-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Knee Dislocations; Multiple Ligament Knee Injuries
Keywords: Knee Injury; Knee Injuries; Knee Surgery; Rehabilitation; Knee Dislocation; Multiple Ligament Knee Injury
MeSH Terms: conditions — Knee Dislocation; Knee Injuries

STUDY DESIGN:
Intervention Model Description: Two parallel prospective randomized multi-center clinical trials. Trial 1 will evaluate the effects of both the timing of surgery and post-operative rehabilitation. Trial 2 will evaluate only the effects of timing of post-operative rehabilitation.
Masking Description: These are unblinded trials as the participants will know when they are receiving surgery and when they are receiving rehabilitation. The data that are collected as part of the standard of care clinical follow-up will be recorded by the clinicians that know the participant's surgery assignment. The primary outcome and most of the secondary outcomes are patient self-report. Given that our interventions are either early or delayed surgery and/or rehabilitation, it is difficult for us to estimate the direction of potential bias (if any) that could come from the unblinded nature of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Early Surgery & Early Rehab (Experimental): Individuals with a MLKI that present within 6 weeks of injury will be randomized to early surgery and early rehabilitation.
  Interventions: Procedure: Early Surgery; Procedure: Early Rehab
- Early Surgery & Delayed Rehab (Experimental): Individuals with a MLKI that present within 6 weeks of injury will be randomized to early surgery and delayed rehabilitation.
  Interventions: Procedure: Early Surgery; Procedure: Delayed Rehab
- Delayed Surgery & Early Rehab (Experimental): Individuals with a MLKI that present within 6 weeks of injury will be randomized to delayed surgery and early rehabilitation.
  Interventions: Procedure: Delayed Surgery; Procedure: Early Rehab
- Delayed Surgery & Delayed Rehab (Experimental): Individuals with a MLKI that present within 6 weeks of injury will be randomized to delayed surgery and delayed rehabilitation.
  Interventions: Procedure: Delayed Surgery; Procedure: Delayed Rehab
- Early Rehab Only (Experimental): Individuals not eligible for randomization to timing of surgery will be randomized to only early rehabilitation.
  Interventions: Procedure: Early Rehab
- Delayed Rehab Only (Experimental): Individuals not eligible for randomization to timing of surgery will be randomized to only delayed rehabilitation.
  Interventions: Procedure: Delayed Rehab

INTERVENTIONS:
Procedure: Early Surgery — Subjects will undergo surgery within 6 weeks after injury.
  Arms: Early Surgery & Delayed Rehab; Early Surgery & Early Rehab
Procedure: Delayed Surgery — Subjects will undergo surgery 12 to 16 weeks after injury.
  Arms: Delayed Surgery & Delayed Rehab; Delayed Surgery & Early Rehab
Procedure: Early Rehab — Subjects will undergo rehabilitation that will include unrestricted range of motion exercises and use of a weightbearing as tolerated gait starting after the first post-operative visit with the surgeon.
  Arms: Delayed Surgery & Early Rehab; Early Rehab Only; Early Surgery & Early Rehab
Procedure: Delayed Rehab — Subjects will undergo rehabilitation that will include use of a knee brace locked in extension, no range of motion exercises and use of non-weightbearing gait for the first 4 weeks after surgery.
  Arms: Delayed Rehab Only; Delayed Surgery & Delayed Rehab; Early Surgery & Delayed Rehab

SUMMARY:
The purpose of this study is to investigate effects of timing of surgery (early vs. delayed) and timing of post-operative rehabilitation (early vs. delayed) for the treatment of military personnel and civilians that sustain a multiple ligament knee injury. To achieve this overall objective of this project, we will conduct two parallel randomized clinical trials. For the first study we will randomize individuals to timing of surgery and timing of post-operative rehabilitation. We hypothesize that early surgery, early rehabilitation and the combination of early surgery with early rehabilitation will lead to an earlier and more complete return to pre-injury military duty, work and sports and better patient-reported physical function. In the second study, those whose timing of surgery can not be randomized, will be only randomized to early or delayed rehabilitation. For this study, we hypothesize that early rehabilitation will lead to an earlier and more complete return to pre-injury military duty, work and sports activity and better patient-reported physical function.

DETAILED DESCRIPTION:
Background:

Multiple ligament knee injuries (MLKIs) represent a spectrum of injury ranging from disruption of two ligaments to all four major ligaments of the knee. Concomitant injuries may include fractures and injuries to vessels, nerves, tendons, menisci and/or articular cartilage. As such, the treatment of MLKIs creates multiple complex problems fraught with complications such as poor wound healing, arthrofibrosis, neurovascular injuries, persistent pain and instability, and post-traumatic osteoarthritis. Following MLKI, individuals are frequently limited with higher demand activities such as in military training, physical labor and sports. Return to duty after combat-related MLKIs has been reported to be as low as 41% and substantially lower than return to work reported for civilians.

There is controversy related to the optimal timing of surgery and post-operative rehabilitation for the treatment of MLKIs. Early surgical intervention for MLKIs has been advocated, however this may be associated with an increased risk for arthrofibrosis. Conversely, delayed surgery may be associated with persistent instability. The best evidence for timing of rehabilitation is based on evidence following ACL reconstruction, where early post-operative rehabilitation is the current standard of care. However, because of the frequency of soft tissue repair procedures, post-operative rehabilitation after surgery for a MLKI typically involves a period of non-WB and delayed ROM exercises. Due to the lack of evidence for the timing of surgery and post-operative rehabilitation, a large scale trial is needed to optimize the outcomes for these potentially devastating injuries. Therefore, this multicenter clinical trial will investigate the effects of timing of surgery and post-op rehabilitation to optimize return to military duty, work and sports for military personnel and civilians with a MLKI.

Objectives, Aims and Hypothesis:

The overall objective of this project is to investigate the effects of timing of surgery (early vs. delayed) and timing of post-op rehabilitation (early vs. delayed) for treatment of MLKIs. To achieve this objective, we will conduct two parallel randomized clinical trials. The related aims and hypotheses are:

Specific Aim 1 and Hypothesis: Determine the effects of timing of surgery and post-op rehabilitation on time to return to pre-injury level of military duty, work and sports and patient-reported physical function. We hypothesize that early surgery, early rehabilitation and the combination of early surgery with early rehabilitation will lead to an earlier and more complete return to pre-injury military duty, work and sports and better patient-reported physical function.

Specific Aim 2 and Hypothesis: For those individuals whose timing of surgery can not be randomized, determine the effects of timing of rehabilitation on time to return pre-injury level of military duty, work and sports and patient-reported physical function. We hypothesize that early rehabilitation will lead to an earlier and more complete return to pre-injury military duty, work and sports activity and better patient-reported physical function.

Overview of Research Procedures:

Male and female military personnel and civilians between the ages of 16 and 55 with a MLKI without a history of prior knee ligament reconstruction that do not have a vascular injury, poly-trauma or a traumatic brain injury will be eligible to participate. After obtaining informed consent, subjects will undergo a preoperative evaluation, including collection of baseline demographics, activity level, and a physical examination.

To address Aim 1, 392 individuals with a MLKI that present within 6 weeks of injury will be randomized to early (within 6 weeks of injury) or delayed (12 to 16 weeks after injury) surgery and early (WB and unrestricted ROM exercises starting first week after surgery) vs. delayed (knee brace locked in extension, no range of motion exercises and non-weightbearing gait for the first 4 weeks after surgery). To address Aim 2, 298 individuals with a MLKI that present greater than 6 weeks after injury, have an injury that precludes randomization to early or delayed surgery as well as those that refuse surgical randomization will be eligible to participate in the trial that compares only early vs. delayed rehabilitation. Randomization will be stratified by study site and knee ligament injury pattern.

Collection of Baseline Demographics and Activity Level:

Following consent and screening, baseline demographic and pre-injury level of military duty, work and sports participation will be recorded. The demographic information to be recorded includes age, sex, weight, height, body mass index (BMI), marital status, education level, pre-injury military duty, work and sports, smoking history and insurance status.

Military Duty - For military personnel, to measure military duty prior to injury we will record the Military Occupational Specialty Physical Demand Classification and will ask three questions from the Injury Surveillance Survey (ability to perform Annual Physical Fitness Test; Deployability and Specific MOS Duties).

Work Activity - To measure work activity prior to injury, we will use the Cincinnati Occupational Rating Scale. Additionally, we will record the individual's pre-injury employment status (work regular duty full time, work regular duty part-time etc.) and occupation.

Sports Activity and Participation - We will use the Marx Activity Rating Scale to measure the subject's level of sports activity in the year prior to injury. To assess sports participation, we will also record the type (very strenuous, strenuous etc.) and frequency (4-7 times per week, 1-3 times per week etc.) of sports participation as well as the specific sport(s) the individual participated in prior to injury.

Baseline Clinical Examination:

A standard of care baseline clinical examination will be performed by the individual's attending orthopaedic surgery. The examination will include assessment of pain, range of motion (ROM), ligament laxity, sensory and neurovascular status (pulses, sensory & motor nerve function). Additionally, standard of care radiographs and MRI will be reviewed to identify fractures and document the ligament injury. The information from the baseline clinical examination will be used to confirm final eligibility in the surgical and post-operative rehabilitation trial or the post-operative rehabilitation only trial.

Interventions:

Aim 1 - Randomization to Early vs. Delayed Surgery and Post-Operative Rehabilitation - Subjects enrolled in the clinical trial for Aim 1 will be randomized to one of four groups: early surgery/early rehabilitation, early surgery/delayed rehabilitation, delayed surgery/early rehabilitation or delayed surgery/delayed rehabilitation.

Those randomized to early surgery will undergo surgery within six weeks of injury and those that are randomized to delayed surgery will undergo surgery 12 to 16 weeks after injury. In all cases, surgery will be in accordance with the principles of anatomic repair/reconstruction of injured structures in a manner that will allow for early range of motion. Surgical reconstruction with allograft or autograft will be performed for mid-substance tears of the ACL and/or posterior cruciate ligament (PCL). Repair or reconstruction will be performed for injury to the medial collateral ligament (MCL) and the posterolateral corner (PLC) structures (fibular collateral ligament, popliteus tendon, and popliteofibular ligament). Injuries to the biceps femoris tendon or iliotibial band will be addressed as necessary. Medial and lateral meniscus tears will be repaired or debrided at the time of surgery. Neuropraxic nerve injuries will not necessitate early intervention; however, if a neurotmesis injury is discovered on MRI, then early intervention for primary repair, grafting or benign neglect may be warranted. All surgical findings and procedures will be documented on electronic surgical case report forms.

Two post-operative rehabilitation protocols have been created, differing only in the time to begin weightbearing (WB) and ROM exercises. After surgery, all individuals will be placed in a hinged brace that is locked in extension. Individuals randomized to early rehabilitation will begin WB as tolerated (WBAT) with the brace locked in full extension and unrestricted ROM approximately 1 week after surgery at the time of the first post-operative visit. Individuals in this group will unlock the brace for ROM exercises, but will keep the brace locked at all other times until the criteria to unlock the brace are met. Weightbearing will be gradually progressed to full WB no earlier than 3 weeks after surgery pending achievement of the criteria for doing so.

Those allocated to delayed rehabilitation will be placed in a knee brace locked in extension, with no range of motion exercise and will utilize a non-weightbearing gait for the first 4 weeks after surgery.

Immediately after surgery both groups will begin isometric quadriceps exercises with the knee in full extension (quad sets, straight leg raises) and high intensity neuromuscular electrical stimulation (NMES) for the quadriceps will be utilized. Use of the post-op brace will be discontinued no earlier than 6 weeks after surgery pending achievement of the criteria to do so. In the Motor Control and Functional Optimization phases of rehabilitation, progression to increasingly demanding activities will be time- and criterion-based to ensure that the individual is advanced safely to reduce the risk of further injury.

Aim 2 - Randomization to only Early vs. Delayed Rehabilitation - Subjects enrolled in the trial for Aim 2 will undergo anatomic surgical repair/reconstruction of the injured structures as described above, however the timing of surgery will be determined by the surgeon and patient after consideration of the individual's specific circumstances related to the nature and extent of the MLKI, associated injuries and timing of presentation. Following surgery, individuals will be randomized to undergo either early or delayed rehabilitation as described above.

Clinical Follow-Up Visits:

Information gathered during standard of care clinical follow-up visits will be prospectively collected at 1 week and 1, 3, 6 and 9 to 12 months after the date of surgery. This information will be documented and will serve to provide additional outcomes related to post-operative recovery. The information will include pain, pain medication usage, joint effusion, wound and neurovascular status, ROM, WB status, use of a post-op rehabilitation brace, imaging and/or laboratory tests ordered and completed, complications and adverse events, additional surgical procedures and military duty, work and sports status. Knee laxity will also be assessed 3, 6 and 9 to 12 months after surgery.

Research Follow-Up Visits:

Subjects in all studies will be followed for 24 months. The primary outcome will be time to return to pre-injury military duty, work and sports. To precisely determine the time to return to military duty, work and sports, we will administer a brief Return to Activity Monitoring Survey on a monthly basis starting 6 months after randomization and continuing through the 24-month follow-up. Patient-reported physical function as measured with the Activity Limitation Scale of the Multiple Ligament Quality of Life (MLQoL) Questionnaire will serve as a co-primary outcome and will be assessed 6, 12 and 24 months after randomization. Secondary outcome measures will include additional knee-specific and general patient-reported measures of physical function and health-related quality of life. We will also collect measures of kinesiophobia, resiliency and functional comorbidities because these constructs may affect return to military duty, work and sports.

ELIGIBILITY:
For the clinical trials for both aims, male and female military personnel and civilians between the ages of 16 and 55 with a MLKI (defined as a complete grade III injury of two or more ligaments) will be eligible to participate. Individuals with a nerve injury or biceps or popliteus tendon rupture or avulsion will not be excluded from participation in either trial.

Individuals will be excluded from both trials if they:

1. Prior knee ligament surgery of the involved knee;
2. Torn or avulsed patellar or quadriceps tendon;
3. Periarticular or long bone fracture that is anticipated to preclude weight-bearing after surgery;
4. Require use of an external fixator for greater than 10 days;
5. Planned staged surgical treatment;
6. Unable to weight bear on the contralateral uninjured leg;
7. Traumatic brain injury (TBI) that limits their ability to participate in their post-operative care;
8. Surgical procedures that precludes early weight-bearing or range of motion.
9. Any condition that would preclude the ability to comply with post-operative guidelines.

Additional Eligibility Criteria for Participation in Aim 1 - Randomization to Both Timing of Surgery and Post-Operative Rehabilitation

To be eligible to participate in the study for Aim 1 individuals with a MLKI must present to orthopaedic surgery in time to undergo definitive surgery within 6 weeks of injury if randomized to the early surgery group.

Individuals will also be ineligible to participate in the study for Aim 1 if they have:

1. Vascular injury that dictates timing of surgery;
2. Poly trauma that precludes surgery within 6 weeks of injury;
3. Skin or soft tissue injury that precludes early surgery and rehabilitation.

Additional Eligibility Criteria for Participation in Aim 2 - Randomization to Only timing of Post-operative Rehabilitation

Subjects with a MLKI that present to orthopaedic surgery at a time that precludes randomization to early surgery or have an injury that precludes randomizing the timing of surgery (such as a vascular injury) as well as those that refuse randomization to the timing of surgery will be eligible to participate in the study for Aim 2 which randomizes subjects to only early vs. delayed rehabilitation.

Individuals will also be excluded from the trial that randomizes only the timing post-operative rehabilitation if they have:

1. Vascular surgery that precludes early rehabilitation;
2. Polytrauma that limits ability to participate in post-operative care;
3. Skin or soft tissue injury that precludes early rehabilitation

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 690 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Time to Return to Pre-Injury Level of Activity | Monthly starting at 6 months post-randomization and continuing to 24 months
  Time to return to pre-injury level military duty, work and/ sports
Patient-Reported Physical Function - Activity Limitation Scale of the Multiple Ligament Quality of Life (MLQoL) Questionnaire | 24 months following randomization
  Activity Limitation Scale of the Multiple Ligament Quality of Life scale measures the degree of difficulty an individual with a multiple ligament knee injury experiences with simple and complex activities as related to his/her knee. The Activity Limitation Scale score ranges from 0 to 100 with a score of 0 representing no activity limitations due to the multiple ligament knee injury.

SECONDARY OUTCOMES:
Physical Impairment Scale of the Multiple Ligament Quality of Life (MLQoL) Questionnaire. | 24 months following randomization
  Physical Impairment Scale measures the physical symptoms experienced by an individual with a multiple ligament knee injury. The Physical Impairment Scale score ranges from 0 to 100 with a score of 0 representing no physical symptoms due to the multiple ligament knee injury.
Emotional Impairment Scale of the Multiple Ligament Quality of Life (MLQoL) Questionnaire | 24 months following randomization
  Emotional Impairment Scale measures the changes in mood and emotions experienced by an individual with a multiple ligament knee injury. The Emotional Impairment Scale score ranges from 0 to 100 with a score of 0 representing no changes in mood and emotions due to the multiple ligament knee injury.
Social Involvement Scale of the Multiple Ligament Quality of Life (MLQoL) Questionnaire | 24 months following randomization
  Social Involvement Scale measures the social limitations experienced by an individual with a multiple ligament knee injury. The Social Involvement Scale score ranges from 0 to 100 with a score of 0 representing no social limitations due to the multiple ligament knee injury.
International Knee Documentation Committee Subjective Knee Form (IKDC-SKF) | 24 months following randomization
  The International Knee Documentation Committee Subjective Knee Form is an 18-item knee-specific patient-reported measure of symptoms, function and sports activities for individuals with a variety of knee conditions, including MLKIs. The International Knee Documentation Committee Subjective Knee Form score ranges from 0 to 100 with higher scores indicating the absence of symptoms and higher levels of function and sports activity.
Patient Reported Outcome Measurement Information System (PROMIS) Physical Function (PF) Scale | 24 months following randomization
  Patient Reported Outcome Measurement Information System Physical Function Scale consists of an item bank of 121 items that assesses physical function regardless of the health condition present that can be administered as a computer adaptive test (CAT) or through the use of short forms. The Physical Function scale scores transformed to a T-score in which a score of 50 represents the US population average with a standard deviation of 10 indicating the population standard deviation.
Patient Reported Outcome Measurement Information System (PROMIS) Global 1- Global 10 | 24 months following randomization
  The Patient Reported Outcome Measurement Information System (PROMIS) Global 10 is a 10-item patient-reported measure of physical and emotional health. The items are combined into two scores, one representing global physical function, the other representing global mental function. The Physical and Emotional Function scores are scores transformed to a T-score in which a score of 50 represents the US population average with a standard deviation of 10 indicating the population standard deviation.
Patient Acceptable Symptom State (PASS) | 24 months following randomization
  The Patient Acceptable Symptom State is a single question that measures an individual's satisfaction with the state of their knee health. The Patient Acceptable Symptom State question is answered Yes or No. A response of Yes indicates that the individual is satisfied with his/her current symptom state.
Global Rating of Change (GRC) | 24 months following randomization
  The Global Rating of Change asks the individual to compare his/her current functional status to his/her functional status at the time of enrollment/post-injury. The responses for the Global Rating of Change range from +7 (greatly better) to -7 (greatly worse). Higher scores representing greater improvement in function since the time of enrollment/post-injury.

CONTACTS AND LOCATIONS:
Overall Officials: James Irrgang, PT, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A public-use version of the dataset will be constructed by the DCC with contents to be determined jointly by the study PIs and the DCC Director. Copies of the public-use version of the dataset will be housed at the DCC on a secure server along with suitable documentation of this dataset. The public-use version of the dataset will be exported by CRF in one or more files in simple, widely-accessible formats, e.g., .xls, .csv, and/or SAS datasets. Documentation will be in .pdf files.
Supporting Information: Study Protocol
Time Frame: The public-use version of the database will be made available 2 years after the study's main paper is published.
Access Criteria: Outside investigators wishing to conduct analyses using the data will submit a request with objectives, methods, and analysis plan to the PI and the Director of the DCC. Once the request is approved, the public-use version of the dataset, with documentation, will be sent by secure email using e-mail, ftp, or other mutually agreeable transmission method.

REFERENCES:
- [Derived] Schenck RC Jr. CORR Insights(R): Is There a Disadvantage to Early Physical Therapy After Multiligament Surgery for Knee Dislocation? A Pilot Randomized Clinical Trial. Clin Orthop Relat Res. 2021 Aug 1;479(8):1737-1739. doi: 10.1097/CORR.0000000000001785. No abstract available. PMID 33944810

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT03543098/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03543098/ICF_001.pdf